CLINICAL TRIAL: NCT05865080
Title: Effect of Intravenous Ketamine Infusion for Hemodynamic Stability in Patients Undergoing Cesarean Delivery
Brief Title: Effect of Intravenous Ketamine Infusion for Hemodynamic Stability in Patients Undergoing Caesarean Delivery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, mohamed, assisstant professor of anesthesia, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 12345
Record Dates: First submitted 2023-04-18; First posted 2023-05-18 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Hemodynamic Instability
Keywords: spinal anesthesia; obstetric anesthesia
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group K (Active Comparator): group K (63 patients): Received 0.3 mg/kg of ketamine IV diluted to 10 ml followed by infusion 0.1 mg/kg/hr. as 20 ml solution,
  Interventions: Drug: Ketamine
- group C (Placebo Comparator): group C (Controlled) (63 patients): Received 10 ml of normal saline followed by infusion of 0.1 ml/kg/hr. as 20 ml solution.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — 0.3 mg/kg of ketamine IV diluted to 10 ml followed by infusion 0.1 mg/kg/hr. as 20 ml solution before spinal anesthesia
  Arms: group K
Drug: Placebo — Normal saline
  Arms: group C

SUMMARY:
Hypotension is the most frequent side effect of intrathecal anesthesia, with a found incidence of more than 80%. With a frequency of between 40% and 60% in patients undergoing surgery, Perioperative shivering is a serious consequence that frequently follows neuraxial anesthesia. This study aimed to determine the multiple advantages of intravenous minimal dose ketamine for intrathecal anesthesia in patients undergoing cesarean delivery

DETAILED DESCRIPTION:
126 female patients undergoing cesarean deliveries, ASA-(II and III) and 21-40 ys old selected from an attendee of outpatient clinics of the Anesthesia Department. Two groups of patients were random to group K (63 patients): Received 0.3 mg/kg of ketamine IV diluted to 10 ml followed by infusion 0.1 mg/kg/hr. as 20 ml solution, group C (Controlled) (63 patients): Received 10 ml of normal saline followed by infusion of 0.1 ml/kg/hr. as 20 ml solution.

ELIGIBILITY:
Inclusion Criter

1. Female patients and full-term,
2. aged between (21 and 40) y. Old.
3. (ASA)-II or III, and undergoing a cesarean section.

Exclusion criteria:

1. Twins and preterm birth.
2. Hypertensive patients and preeclamptic patients.
3. Morbidly obese patients.
4. Spinal anesthesia contraindication as the patient refused, severe mitral or tricuspid stenosis and local sepsis.

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Hemodynamics | Up to 24 hours after operation
  Primary outcomes: Hemodynamic parameters (MAP and HR). Secondary outcomes
  1. Incidence of intraoperative shivering.
  2. The postoperative pain was assessed by VAS score.
  3. Sedation score in between groups.
  4. Fetus evaluated by Apgar score.
  5. Postoperative side effects as nausea, vomiting, nystagmus, diplopia, and hallucinations.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine -Al-Azhar university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided